CLINICAL TRIAL: NCT07010796
Title: Treatment of Adipose Tissue and Skin Laxity at the Buttocks by PDLLA, US and RF
Status: Completed | Type: Observational
Sponsor: Pablo Naranjo García, MD (Other)
Responsible Party: Sponsor-Investigator, Pablo Naranjo García, MD, Principle Investigator Pablo Naranjo Garcia, MD, Elite Laser Clinic
Organization: Elite Laser Clinic (Other)
Other Study IDs: PDLLA-UD/RF-01
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Local Fat Deposits

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Alma Prime X — Alma Prime x is a platform that provides applicators for radiofrequency and ultrasound.

SUMMARY:
Local body fat and lax skin is treated with a combined approach of PDLLA injections and topical ultrasound and radiofrequency.

ELIGIBILITY:
Inclusion Criteria:

* adults over 18 years
* patients eligible to be treated with radiofrequency and ultrasound
* all genders

Exclusion Criteria:

* patients displaying contraindications for treatment with radiofrequency and ultrasound
* pregnancy
* immune diseases
* active virus infections

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants were selected due to their desire to reduce fat deposits at the buttock area as well as tightening lax skin.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
change of fat deposits | From enrollment to the end of treatment at 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Elite Laser Clinic Organization, Madrid, Spain